CLINICAL TRIAL: NCT03521427
Title: Effects of Intensive Upper and Lower Limbs Motor Control Therapy in Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Collaborators: European University Spain (Other)
Responsible Party: Principal Investigator, Isabel Rodriguez Costa, PhD, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-0066/16
Record Dates: First submitted 2017-06-29; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cerebral Palsy
Keywords: Intensive Therapy; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive bimanual therapy (Experimental): Ninety hours of intensive bimanual therapy
  Interventions: Other: Intensive bimanual therapy
- Neurodevelopmental treatment (Active Comparator): Ninety hours of intensive neurodevelopmental therapy
  Interventions: Other: Intensive neurodevelopmental therapy

INTERVENTIONS:
Other: Intensive bimanual therapy — Ninety hours of intensive bimanual therapy
  Arms: Intensive bimanual therapy
Other: Intensive neurodevelopmental therapy — Ninety hours of intensive neurodevelopmental therapy
  Arms: Neurodevelopmental treatment

SUMMARY:
The aim of the study is to determine the effetiveness of the intensive upper and lower limbs therapy to improve the funtional outcomes and to minimize ther energetic spendings during funtional activities in Cerebral Palsy patients.

DETAILED DESCRIPTION:
The aim of the study is to determine the effetiveness of the intensive upper and lower limbs therapy to improve the funtional outcomes and to minimize ther energetic spendings during funtional activities in Cerebral Palsy patients. Also to know paretns and caregivers perceptions.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy

Exclusion Criteria:

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2018-02-03 (Actual)

PRIMARY OUTCOMES:
Arm Funtion | 6 months
  Assissting Hand Assessment Instrument (AHA)

SECONDARY OUTCOMES:
Funtional Activity | 6 months
  Jebsen Taylor Hand Funtion Test
Perception of performance in everyday living | 6 months
  Canadian Occupational Performance Measure (COMP)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gordon, PhD, Study Director — Columbia Universuty
Locations (1):
- University, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No